CLINICAL TRIAL: NCT05890963
Title: Phase 1b Single Dose Clinical Trial of a Novel Long-Acting Bispecific Antibody in People With HIV to Inform Development for HIV Pre- and Post-Exposure Prophylaxis
Brief Title: 10E8.4/iMab Bispecific Antibody and VRC07-523LS Monoclonal Antibody in HIV-infected Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Ho (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); US Military HIV Research Program (Network); National Institute of Allergy and infectious Diseases (NIAID)/Vaccine Research Center (VRC) (Unknown)
Responsible Party: Sponsor-Investigator, David Ho, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAU5207; W81XWH-18-2-0040 (Other Grant/Funding Number: U.S. Military HIV Research Program (MHRP)); RV584 (Other: WRAIR IRB)
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: HIV-1-infection
Keywords: Antiretroviral therapy (ART); VRC07-523LS; 10E8.4/iMab; Monoclonal antibody; Bispecific antibody; Broadly neutralizing antibodies; Viral suppression; Ibalizumab; 10E8
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active; ibalizumab

STUDY DESIGN:
Intervention Model Description: Participants are assigned to 1 to 5 arm sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: Oral ART (Active Comparator): Participants will receive standard daily oral ART.
  Interventions: Drug: ART
- Arm 2: 10E8.4/iMab 600mg IV. (Experimental): Participants will receive a single dose of 10E8.4/iMab 600mg IV.
  Interventions: Drug: 10E8.4/iMab
- Arm 3: 10E8.4/iMab 600mg IM. (Experimental): Participants will receive a single dose of 10E8.4/iMab 600mg IM.
  Interventions: Drug: 10E8.4/iMab
- Arm 4:10E8.4/iMab 1800mg IV. (Experimental): Participants will receive a single dose of 10E8.4/iMab 1800mg IV.
  Interventions: Drug: 10E8.4/iMab
- Arm 5: Combination 10E8.4/iMab and VRC07-523LS therapy (Experimental): Participants will receive a single dose of combination therapy with both 10E8.4/iMab 1800mg IV. and VRC07-523LS 1200mg IV.
  Interventions: Drug: 10E8.4/iMab; Drug: VRC07-523LS

INTERVENTIONS:
Drug: ART — ART is a combination of three or more drugs from different classes of antiretroviral medication.
  Other Names: antiretroviral therapy
  Arms: Arm 1: Oral ART
Drug: 10E8.4/iMab — 10E8.4/iMab is an engineered bispecific antibody with two arms combined into a single molecule that exhibits synergistic enhancement of antiviral activity. 10E8.4/iMab will be administered IV at the 600mg or 1800mg dose or IM at 600mg dose to participants in Step 1 per the Schedule of Events (SOE) based on the arm the participant is assigned.
  Other Names: ibalizumab
  Arms: Arm 2: 10E8.4/iMab 600mg IV.; Arm 3: 10E8.4/iMab 600mg IM.; Arm 4:10E8.4/iMab 1800mg IV.; Arm 5: Combination 10E8.4/iMab and VRC07-523LS therapy
Drug: VRC07-523LS — VRC07-523LS is an engineered variant of VRC01, a bNAb that targets the CD4 binding site of the HIV-1 envelope. VRC07-523LS will be administered IV at the 1200mg dose to participants in Step 1 per the SOE.
  Other Names: VRC01 variant
  Arms: Arm 5: Combination 10E8.4/iMab and VRC07-523LS therapy

SUMMARY:
This is an open-label phase 1b clinical trial enrolling people living with HIV (PLWH) who are antiretroviral therapy (ART)-naïve or have not been on ART for > 24 weeks. This study will enroll PLWH to assess the safety, tolerability, and antiviral effect of bispecific and long-acting bNAbs, alone and in combination. The study will be conducted as a single center study at National Institute for Medical Research-Mbeya Medical Research Center (NIMR-MMRC) in Mbeya, Tanzania.

20 PLWH will be sequentially enrolled into one of 5 arms, each arm comprised of 4 participants. Sequential enrollment will occur in the following order:

* Arm 1 will receive standard daily oral ART.
* Arm 2 will receive a single dose of 10E8.4/iMab 600mg intravenous injection (IV).
* Arm 3 will receive a single dose of 10E8.4/iMab 600mg intramuscular injection (IM).
* Arm 4 will receive a single dose of 10E8.4/iMab 1800mg IV.
* Arm 5 will receive a single dose of combination therapy with both 10E8.4/iMab 1800mg IV and VRC07-523LS 1200mg IV.

DETAILED DESCRIPTION:
Although global initiatives have made great strides in controlling the human immunodeficiency virus (HIV) pandemic, HIV and acquired immune deficiency syndrome (AIDS) continue to impact the lives and livelihoods of a significant portion of the population. In 2019, 38 million individuals were living with HIV and 690,000 died of AIDS-related causes. Despite extensive global efforts for disease control over the last 20 years, 1.7 million individuals contract HIV annually. Antiretroviral therapy (ART) reduces morbidity and mortality associated with HIV by suppressing viral replication but does not eradicate infection. There are barriers to universal ART use that include toxicities, costs, drug resistance, and the need for lifelong adherence. To overcome these barriers, HIV broadly neutralizing antibodies (bNAbs) represent a novel approach to HIV prevention and treatment.

The primary endpoint of change in viral load will be assessed at day 14. Participants will then transition to Step 2, during which all participants will take standard daily oral ART and have viral load monitored through Step 2 week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write in Kiswahili and/or English
2. Able and willing to provide written informed consent
3. Passes Test of Understanding (TOU)
4. Aged 18-50 years, inclusive
5. Antiretroviral Therapy (ART)-naïve or no ART for > 24 weeks at the time of screening
6. HIV RNA 1,000-100,000 copies/mL
7. CD4 ≥ 500 cells/mm3
8. Laboratory criteria at screening within protocol-specified limits for blood, chemistry and urinalysis
9. Willing and able to participate in study visits and procedures for up to 50 weeks
10. Willing and able to begin ART as directed during the study
11. Willing and able to use barrier protection during sex with partners without HIV or partners with unknown HIV status throughout Step 1 and until viral suppression <200 copies/mL is confirmed in Step 2
12. Willing and able to adhere to the following contraception requirements:

    1. Participants who are able to become pregnant must agree to use at least one method of highly effective contraception if participating in sexual activity that could lead to pregnancy. This must begin at least 14 days prior to study enrollment.
    2. Participants who engage in sexual activity that could lead to their partner becoming pregnant and who are of reproductive potential must agree to use a barrier method of contraception to avoid pregnancy in a sexual partner of reproductive potential. The barrier method must be used for the duration of the study.

Exclusion Criteria:

1. Weight >100 kg
2. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational (other than for the prevention and/or treatment of SARS-CoV2/COVID-19)
3. History of viral failure on two or more ART regimens
4. Planned or anticipated need for enfuvirtide, maraviroc, fostemsavir, or ibalizumab for antiretroviral therapy.
5. AIDS-defining illness, as enumerated by the WHO Stage 3 or 4, within the six months prior to enrollment
6. Ongoing oral thrush
7. Active injection or other recreational drug use within the previous 12 months that, in the opinion of the investigator, would impede the participant's ability to safely and consistently adhere to the study protocol
8. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment.
9. History of chronic urticaria requiring daily treatment
10. Known active hepatitis B virus infection or positive hepatitis B surface antigen at any time in the past
11. Known active hepatitis C virus infection or positive hepatitis C antibody at any time in the past
12. Untreated syphilis
13. Estimated GFR < 50 mL/min within the past 90 days
14. Pregnant or breast-feeding
15. Receipt of licensed vaccine or other investigational study agent within 28 days prior to enrollment or any past participation in an investigational HIV vaccine study with receipt of active product
16. Current or planned participation in another interventional clinical trial during the study period, including clinical trials of investigational new drugs or investigating a new application for an approved medication
17. Chronic or recurrent use of medications that modify host immune response, such as oral steroids, parenteral steroids, or cancer chemotherapy (note: locally-acting medications-such as inhaled, topical, or intra-articular steroids-are allowed)
18. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the participant including, but not limited to: diabetes mellitus type I, chronic hepatitis, renal failure; OR clinically significant forms of: drug or alcohol abuse, mental illness, severe asthma, autoimmune disease, decompensated psychiatric disorders, hypertension, heart disease, or cancer
19. Any medications that, in the opinion of the investigator, would preclude intramuscular injections
20. Study site employee

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Grade 3 or higher antibody-related reactogenicity and adverse events | Up to Week 48 in Step 2
  Includes potentially life-threatening, or fatal events.
Change in plasma HIV RNA from day 0 to day 14 | Day 0 and Day 14 in Step 1
  Viral RNA copies/mL will be measured.
Proportion of participants with HIV RNA < 50 copies/mL at day 14 | Up to Day 14 in Step 1
  Percentage of participants will be calculated.

SECONDARY OUTCOMES:
Proportions of participants with HIV RNA <50 copies/mL | Up to Week 48 in Step 2
  Percentage of participants will be calculated.
Proportions of participants with HIV RNA < 200 copies/mL | Up to Week 48 in Step 2
  Percentage of participants will be calculated.
Proportions of participants with HIV RNA <1000 copies/mL | Up to Week 48 in Step 2
  Percentage of participants will be calculated.
Peripheral HIV RNA | Up to Week 48 in Step 2
  Serum level of viral RNA (copies/mL) will be measured.
Plasma level of 10E8.4/iMab | Up to Week 48 in Step 2
  Serum level of 10E8.4/iMab (ug/mL) will be measured.
Plasma level of VRC07-523LS | Up to Week 48 in Step 2
  Serum level of VRC07-523LS (ug/mL) will be measured.
CD4 receptor occupancy | Up to Week 48 in Step 2
  The percentage of CD4 cells that bind to 10E8.4/iMab will be measured.
HIV reservoir size | Up to Week 48 in Step 2
  Will measure HIV DNA in copies/million cells.
Neutralization sensitivity of 10E8.4/iMab | Up to Week 48 in Step 2
  Half-maximal inhibitory concentration (IC50) will be measured.
Neutralization sensitivity of VRC07-523LS | Up to Week 48 in Step 2
  Half-maximal inhibitory concentration (IC50) will be measured.
Presence of anti-bNAb antibodies | Up to Week 48 in Step 2
  The anti-drug antibody titer in serum will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Missanga, MD, Principal Investigator — NIMR-MMRC; David D. Ho, MD, Principal Investigator — Columbia University Irving Medical Center (IND Sponsor); Trevor A. Crowell, MD, PhD, Study Chair — The U.S. Military HIV Research Program (MHRP)
Locations (1):
- National Institute for Medical Research-Mbeya Medical Resarch Center, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results published in any manuscript or otherwise disseminated will be shared. Sharing would occur only after deidentification and with researchers who provide a methodologically sound proposal to analyze the data and secure required regulatory and ethical approvals through appropriate institutions. Deidentified data may also be made available through public data repositories.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the study.
Access Criteria: Data will only be shared with proper approvals in place to entities that are approved to access the data according to the sponsor.

REFERENCES:
- [Background] Huang Y, Yu J, Lanzi A, Yao X, Andrews CD, Tsai L, Gajjar MR, Sun M, Seaman MS, Padte NN, Ho DD. Engineered Bispecific Antibodies with Exquisite HIV-1-Neutralizing Activity. Cell. 2016 Jun 16;165(7):1621-1631. doi: 10.1016/j.cell.2016.05.024. PMID 27315479
- [Background] Mahomed S, Garrett N, Capparelli EV, Osman F, Harkoo I, Yende-Zuma N, Gengiah TN, Archary D, Samsunder N, Baxter C, Mkhize NN, Modise T, Carlton K, McDermott A, Moore PL, Karim QA, Barouch DH, Fast PE, Mascola JR, Ledgerwood JE, Morris L, Abdool Karim SS. Safety and Pharmacokinetics of Monoclonal Antibodies VRC07-523LS and PGT121 Administered Subcutaneously for Human Immunodeficiency Virus Prevention. J Infect Dis. 2022 Aug 26;226(3):510-520. doi: 10.1093/infdis/jiac041. PMID 35134995
- [Background] Huang J, Ofek G, Laub L, Louder MK, Doria-Rose NA, Longo NS, Imamichi H, Bailer RT, Chakrabarti B, Sharma SK, Alam SM, Wang T, Yang Y, Zhang B, Migueles SA, Wyatt R, Haynes BF, Kwong PD, Mascola JR, Connors M. Broad and potent neutralization of HIV-1 by a gp41-specific human antibody. Nature. 2012 Nov 15;491(7424):406-12. doi: 10.1038/nature11544. Epub 2012 Sep 18. PMID 23151583
- [Background] Burkly LC, Olson D, Shapiro R, Winkler G, Rosa JJ, Thomas DW, Williams C, Chisholm P. Inhibition of HIV infection by a novel CD4 domain 2-specific monoclonal antibody. Dissecting the basis for its inhibitory effect on HIV-induced cell fusion. J Immunol. 1992 Sep 1;149(5):1779-87. PMID 1380539
- [Background] Jacobson JM, Kuritzkes DR, Godofsky E, DeJesus E, Larson JA, Weinheimer SP, Lewis ST. Safety, pharmacokinetics, and antiretroviral activity of multiple doses of ibalizumab (formerly TNX-355), an anti-CD4 monoclonal antibody, in human immunodeficiency virus type 1-infected adults. Antimicrob Agents Chemother. 2009 Feb;53(2):450-7. doi: 10.1128/AAC.00942-08. Epub 2008 Nov 17. PMID 19015347
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Wolfe D, Carrieri MP, Shepard D. Treatment and care for injecting drug users with HIV infection: a review of barriers and ways forward. Lancet. 2010 Jul 31;376(9738):355-66. doi: 10.1016/S0140-6736(10)60832-X. PMID 20650513
- [Background] Jaworski JP, Cahn P. Preventive and therapeutic features of broadly neutralising monoclonal antibodies against HIV-1. Lancet HIV. 2018 Dec;5(12):e723-e731. doi: 10.1016/S2352-3018(18)30174-7. Epub 2018 Sep 21. PMID 30245003
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822